CLINICAL TRIAL: NCT03088371
Title: Psoas Sciatic Blockade Could be a Sole Anaesthetic Technique for Total Knee Arthroplasty
Brief Title: Psoas Sciatic Blockade for Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Dr Ezzeldin Ibrahim, Assistant Professor in anaesthesia, intensive care, and pain medicine., Menoufia University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: MenoufiaU2017
Record Dates: First submitted 2017-03-13; First posted 2017-03-23 (Actual); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Knee Osteoarthritis
Keywords: Total knee replacement; Psoas Sciatic block; Epidural anaesthesia
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Bupivacaine; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psoas Sciatic blockade (Other): Psoas Sciatic blockade with 20 ml lidocaine 1% and 20 ml bupivacaine 0.25% pajunk needle used for the block and 5 ml Lidocaine 2% used for post-operative pain.
  Interventions: Drug: Bupivacaine 0.25%; Other: Pajunk Needle; Drug: Lidocaine 1%; Drug: Lidocaine 2 %
- Combined spinal epidural (Other): Spinal anaesthesia with 2.5 ml (12.5 mg) of heavy Bupivacaine 0.5%. Epidural for post-operative pain with Bupivacaine 0.125 %in a rate of 7-10 ml/hour Portex combined spinal epidural kit needle through needle.
  Interventions: Other: Portex combined spinal epidural kit; Drug: Bupivacaine 0.5%; Drug: Lidocaine 2 %; Drug: Bupivacaine 0.125 %

INTERVENTIONS:
Drug: Bupivacaine 0.25% — For psoas sciatic block.
  Other Names: Bupivacaine
  Arms: Psoas Sciatic blockade
Other: Pajunk Needle — For local anaesthesia application in psoas sciatic block
  Arms: Psoas Sciatic blockade
Other: Portex combined spinal epidural kit — For combined spinal epidural anaesthesia
  Arms: Combined spinal epidural
Drug: Lidocaine 1% — For psoas sciatic block.
  Other Names: Lidocaine
  Arms: Psoas Sciatic blockade
Drug: Bupivacaine 0.5% — For spinal anaesthesia in combined spinal epidural anaesthesia.
  Other Names: Bupivacaine
  Arms: Combined spinal epidural
Drug: Lidocaine 2 % — For psoas sciatic block in the post-operative period
  Other Names: Lidocaine
Drug: Bupivacaine 0.125 % — For combined spinal epidural in the post-operative period.
  Other Names: Bupivacaine
  Arms: Combined spinal epidural

SUMMARY:
Objectives: To compare the efficacy of continuous combined psoas sciatic block as a sole anaesthetic technique with conventional combined spinal epidural anesthesia for patients undergoing total knee arthroplasty.

Subjects and Method: Eighty patients ASA (American society of anaesthesiologists classification) I to III with age range from 50 to 65 years old and scheduled for total knee replacement were included in the study. Subjects were divided into two groups; the first group (Pso/sci) received ultrasound guided with the use of nerve locator continuous psoas sciatic block and the second group (CSE) received combined spinal epidural anesthesia. Onset of sensory and motor block time, hemodynamic changes, contra-lateral spread, first time need for analgesia, incidence of complications, and patient and surgeon satisfactions were recorded.

DETAILED DESCRIPTION:
After approval of the ethics committee, department of anaesthesia, Menoufia university and written informed consent, 80 patients undergoing unilateral total knee arthroplasty were randomly allocated into two groups. The first group (40 patients) received continuous psoas compartment block combined with continuous sciatic block (Pso/Sci group) and the second group (40 patients) received combined spinal epidural anaesthesia (CSE group). All patients were between 50 and 65 years old with an American society of anaesthesiologists classification (ASA status) of I to III. Patients' exclusion criteria included contraindication of regional anesthesia, bleeding disorders, localized infection, neurological deficit, substance dependence, and uncooperative patients. Upon arrival to the operative theater patients were attached to the standard monitoring and an intravenous cannula was inserted. All patients received 1 - 2 mg midazolam for sedation before the blocks.

Sciatic nerve blockade:

The block was done under complete aseptic technique. The patient was positioned in the lateral recumbent position with the operative side up and the hips and knees were flexed. The greater trochanter, posterior superior iliac spine and sacral hiatus were palpated and marked. Curvilinear low frequency U/S probe 2-5 MHz, (Sonosite, M-Turbo, Sonosite Inc., USA) was used for scanning. The probe was placed transversely in the middle of the line connecting the greater trochanter and sacral hiatus. The hip joint and the ischial spine were seen as hyperechoic lines in the lateral and medial sides respectively and the sciatic nerve was appeared as a triangular or flattened hyperechoic structure under the gluteus maximus. Local infiltration with 1 ml lidocaine 2% with 27-gauge needle was done before introducing the 100 mm 18 gauge sterile insulating pajunk needle (PAJUNK, PlexoLong, Germany) for the block.

The pajunk needle was connected to a nerve stimulator (Plexygon, Vygon Italia, Padua, Italy) with 0.8 mA initial current and inserted out of plane reaching the sciatic nerve until eliciting either planter flexion or dorsiflexion with reduced current output up to 0.2 mA. A mixture of 15 ml lidocaine 1% and 15 ml bupivacaine 0.25% were injected around the sciatic nerve. A multi-perforated reinforced catheter was inserted through the needle and advanced 5 cm distal to the needle tip to provide continuous infusion. The needle was removed and the catheter was fixed to the skin.

Psoas compartment blockade:

The block was done under complete aseptic technique. The patient was positioned in the lateral recumbent position with the operative side upper most and hip and knee were flexed. L4-5 space was identified and marked by a line passing between the iliac crest and vertebral column. The puncture point for the block was marked 5 cm lateral to the L4-5 space within the drawn line. Using curvilinear low frequency U/S probe 2-5 MHz, (Sonosite, M-Turbo, Sonosite Inc., USA) the area was scanned longitudinally starting from the sacrum and moving cranially to identify the 4th transverse process then turned transversally in a rocking manner laterally to the end of the transverse process. The skin at the site of entry was infiltrated with 1 ml lidocaine 2% using 27-gauge needle. A 100 mm 18 gauge insulating pajunk needle (PAJUNK, PlexoLong, Germany) connecting to a nerve stimulator (Plexygon, Vygon Italia, Padua, Italy) with 0.8 mA initial current was advanced from medial to lateral proximal to the transverse process of L4 then advanced caudally to it until eliciting the quadriceps femoris contraction. When the contraction was persisted with reduced current down to 0.2 mA, a mixture of 20 ml lidocaine 1% and 20 ml bupivacaine 0.25% were injected after repeated negative aspiration. A multi-perforated reinforced catheter was inserted through the pajunk needle and was advanced 5 cm distal to the needle tip. The needle was removed and catheter was fixed to the skin.

Combined spinal epidural block:

The patient was in the sitting position, L3-4 space was marked then the area was sterilized and draped. Local anaesthetic (LA) was applied in the track by 27 gauge needle with 5 ml Lidocaine 1%. With portex combined spinal epidural kit needle through needle (PORTEX, Smiths Medical ASD, Inc., USA), the epidural space was detected by loss of resistance technique with saline then 27 gauge 120 mm pencil point spinal needle passed through the epidural needle till perforating the dura and observing the cerebrospinal fluid, 2.5 ml (12.5 mg) of heavy bupivacaine 0.5% (Bupivacaine hydrochloride 0.5%, 5mg/ml, AstraZeneca) was injected. The needle was removed and the epidural catheter was advanced 4 cm distal to the needle tip and fixed to the skin.

After block was done all the patients returned back to the supine position, the sensory block was assessed by cold perception using ice backs and the motor block was assessed by Bromage scale (3=no flexion of hip, knee and foot; 2=no flexion of hip and knee with foot flexion; 1=no flexion of hip with flexion of knee and foot; 0=full flexion of hip, knee and foot). Sensory and motor blocks were assessed every 10 minutes for 3 times. Bilateral assessment was done to detect epidural spread of local anesthetics. Failure to establish adequate sensory and motor blocks after 30 minutes, a failed block was considered and general anesthesia was induced if there were no contraindications and the patient was excluded from the study.

In both groups, the time taken to finish the block was recorded. The onset of sensory and motor blocks were recorded which was defined as the time from finishing the blockade to the occurrence of the block.

In the post-operative period, the duration of the sensory block for both groups was recorded which was defined as the time between the onset of the block and the asking for first analgesia. Once the patient experienced pain (VAS ≥ 3), a bolus of 5 ml Lidocaine 2 % was injected in both catheters in (pso/sci) group and epidural catheter in (CSE) group then continuous LA infusion was followed using a solution of 0.125 % Bupivacaine in a rate of 7-10 ml/hour according to the patient response. Heart rate and blood pressure were recorded every 5 minutes all through the procedures; bradycardia and hypotension were considered if the heart rate and the mean blood pressure were 30% below the starting baseline. Bradycardia was treated by IV 0.5 mg atropine and hypotension was managed by 10- 15 mg IV ephedrine. Intra- and post-operative side effects like bradycardia, hypotension, nausea and vomiting were recorded. Age, gender, weight, ASA class and duration of surgery (time from skin incision until skin closure) were recorded. Data was analyzed using SSPS software 12.0 (SSPS Inc., Chicago, IL, USA) and represented as mean ± standard deviation and p value less than 0.05 was considered to be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing total knee arthroplasty with ASA I, II, or III.

Exclusion Criteria:

* Patients refusal, allergy to drugs used, and uncooperative patients.

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-04-10 (Actual); Primary Completion 2016-06-14 (Actual); Study Completion 2016-09-22 (Actual)

PRIMARY OUTCOMES:
Duration of sensory block | 24 hours post-operative.
  Duration of the sensory block is the time from the onset of the block to the first call of analgesia (minutes).

SECONDARY OUTCOMES:
Mean arterial blood pressure | Intra-operative
  Mean arterial blood pressure (mmHg) was recorded for both groups
Heart rate | Intra-operative.
  Heart rate (beats/minute) was recorded for both groups
Time of mobilisation | 24 hours post-operative.
  Time of mobilisation is the time after admission to the surgical word when the patient can get out of bed for more than 15 minutes with or without support.
Patients' satisfaction questionnaire | Peri-operative
  The patients were asked if they were happy with the procedure or not.
Surgeons' satisfaction questionnaire | Peri-operative
  The surgeons were asked if they were happy with the anaesthetic technique and if it was adequate for the surgical procedure or not.

IPD SHARING:
Plan to Share IPD: No